CLINICAL TRIAL: NCT05755347
Title: Assessing Functional Status Needs Via Patient-Reported Outcomes Measures in the Pre-treatment Setting With Metastatic Breast Cancer Patients
Brief Title: Assessing Functional Status Needs Via PRO Measures for Pts With Metastatic Breast Cancer
Status: Completed | Type: Observational
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: LCCC2241
Record Dates: First submitted 2023-02-22; First posted 2023-03-06 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Breast Cancer; Metastasis
Keywords: patient reported outcomes; quality of life; functional status
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Single Arm: Subjects with metastatic breast carcinoma have been receiving treatment at the study center and responding to survey questionnaires.
  Interventions: Other: General health survey questionnaires; Other: PROMIS Cancer Function Brief 3D profile questionnaires; Other: FACT-G questionnaires; Other: Godin Leisure-Time Exercise Questionnaire; Other: REAP-S questionnaires

INTERVENTIONS:
Other: General health survey questionnaires — Patient-reported outcome survey will be offered at baseline.
Other: PROMIS Cancer Function Brief 3D profile questionnaires — Patient-reported outcome survey will be offered at baseline.
Other: FACT-G questionnaires — Patient-reported outcome survey will be offered at baseline.
Other: Godin Leisure-Time Exercise Questionnaire — Patient-reported outcome survey will be offered at baseline.
Other: REAP-S questionnaires — Patient-reported outcome survey will be offered at baseline.

SUMMARY:
The purpose of this single-site non-randomized study is to identify areas of need related to functional status and overall health, including nutrition and mental health in subjects with metastatic breast cancer (MBC). A decline in functional status is observed after breast cancer diagnosis and exacerbated by treatment. Declining functional status impacts the quality of life and can lead to increased comorbidity burden, hospitalization, and increased mortality. Functional status is assessed by specific provider-graded scales. Patient Reported Outcome (PRO) measures may better assess certain aspects of patient health and symptom domains. Thus, potentially supporting the future implementation of effective prehabilitation strategies. This study explores whether a PRO-based survey will identify the physical and emotional health and the social and financial status of patients newly diagnosed with MBC.

ELIGIBILITY:
In order to participate in this study a subject must meet all of the eligibility criteria outlined below.

Inclusion Criteria:

1. Written informed consent was obtained from participants in the study and HIPAA authorization for release of personal health information.
2. Subject is willing and able to comply with study procedures based on the judgment of the investigator or protocol designee.
3. Age ≥ 18 years at the time of consent.
4. Recent diagnosis of new metastatic breast cancer at time of screening.

Exclusion Criteria:

1. Exclusion Criteria
2. Inability to read or speak English.
3. Dementia, altered mental status, or any psychiatric condition as determined by clinical or study team that would prohibit the understanding or rendering of informed consent.
4. Current incarceration.
5. Subject has already received treatment for metastatic breast cancer prior to screening.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Subject with metastatic breast cancer receive treatment at the University of North Carolina, Lineberger Comprehensive Cancer Center.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2023-03-17 (Actual); Primary Completion 2024-02-05 (Actual); Study Completion 2024-02-05 (Actual)

PRIMARY OUTCOMES:
Physical activity levels | Baseline
  Physical activity levels will be measured using the Godin Leisure-Time Exercise Questionnaire. Godin Leisure-Time Exercise Questionnaire has 3 dichotomous questions, answers will be "yes" or "no". There will be reason questions if the answer is no.

SECONDARY OUTCOMES:
Acceptability of survey | Baseline
  Acceptability of survey to subjects will be measured by the percentage of eligible patients who complete the survey.
Health-related quality of life - FACT-G | Baseline
  Health-related quality of life will be measured by Functional Assessment of Cancer Therapy (FACT-G) which is a survey assessing physical, emotional, and functional well-being on a Likert-type scale. higher scores demonstrating higher health-related quality of life, from 0 to 4. Higher scores represent better QOL.
Health-related quality of life - PROMIS | Baseline
  The patient-Reported Outcomes Measurement Information System (PROMIS) survey will assess physical function, fatigue, and social participation. This survey was designed for cancer rehabilitation needs. It asks patients on a Likert-type scale about their ability to perform mobility and activities of daily living tasks along with the frequency of fatigue and ability to participate in vocational and avocational activities.
Diet quality | Baseline
  The diet quality will be measured using a modified version of the Rapid Eating Assessment for Participants (REAP-S) survey will assess diet and nutrition quality. For the general population, a score of 32 or higher determines a high-quality/desirable diet. The survey asks about the intake of nutrients including vegetables/fruit, whole grains, types of fat, calcium-rich foods, and others. Responses usually/often receive 1 point, sometimes receive 2 points, and rarely/do not apply to receive 3 points.
the percentage of subjects referred | Baseline
  the percentage of subjects referred will be defined as subjects who have been referred to or used Lineberger Comprehensive Cancer Center supportive services for patients Referral rates will be reported for an array of the University of North Carolina Lineberger supportive services by questionnaire.
Barriers to access exercise | Baseline
  Barriers to accessing exercise will be evaluated by questionnaire.
health-related opinions | Baseline
  Health-related opinions regarding prehabilitation interventions will be assessed by questionnaire which includes open-ended questions.

CONTACTS AND LOCATIONS:
Overall Officials: Sasha Knowlton, MD, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (1):
- Lineberger Comphrehensive Cancer Center at University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Clinical trials at UNC Lineberger — http://unclineberger.org/patientcare/clinical-trials/clinical-trials